CLINICAL TRIAL: NCT04052737
Title: A Prospective, Multicentric, Randomized, Double Blind, Placebo Controlled Phase II Clinical Study to Compare the Safety and Efficacy of PMZ-1620 Therapy Along With Standard Supportive Care in Subjects of Mild to Moderate Alzheimer's Disease
Brief Title: PMZ-1620 (Sovateltide) in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-1620/CLINICAL-2.2/2017; CTRI/2017/12/011003 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Endothelin; Neurogenesis; Neural progenitor cells
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — sovateltide

STUDY DESIGN:
Intervention Model Description: In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour (total dose/day: 0.9 µg/kg body weight). The same dosing regimen will be repeated every month for 6 months post randomization.
  In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1 post randomization. The same dosing regimen will be repeated every month for 6 months post randomization.
  In both treatment groups, subjects will be provided the best available standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): Patients will receive the best available standard of care. In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, the same dosing regimen will be repeated every month for 6 months post randomization.
  Interventions: Drug: Normal Saline along with standard treatment
- PMZ-1620 (sovateltide) (Experimental): Patients will receive the best available standard of care. In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1 (total dose/day: 0.9 µg/kg body weight), the same dosing regimen will be repeated every month for 6 months post randomization.
  Interventions: Drug: PMZ-1620 (sovateltide) along with standard treatment

INTERVENTIONS:
Drug: Normal Saline along with standard treatment — PMZ-1620 (sovateltide) is an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in Alzheimer's disease patients. In this arm normal saline along with standard treatment will be given for active comparison.
  Other Names: Vehicle
  Arms: Normal Saline
Drug: PMZ-1620 (sovateltide) along with standard treatment — PMZ-1620 (sovateltide) is an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in Alzheimer's disease patients.
  Other Names: IRL-1620
  Arms: PMZ-1620 (sovateltide)

SUMMARY:
This is a prospective, multicentric, randomized, double blind, placebo controlled Phase II clinical study to compare the safety and efficacy of PMZ-1620 therapy along with standard supportive care in subjects with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's is not just a disease of old age, approximately 200,000 Americans under the age of 65 having younger-onset Alzheimer's disease (AD). In 2015, there were approximately 29.8 million people worldwide with AD. The person with Alzheimer's disease can live an average of eight years after their symptoms become noticeable to others, but survival range is 4 to 20 years, depending on the age and other health conditions (www.alz.org). The pathophysiology of AD is related to the injury and death of neurons, initiating in the hippocampus brain region that is involved with memory and learning, then atrophy affects the entire brain. The cause of Alzheimer's disease is still poorly understood and about 70% of the risk is associated with genetic. Other risk factors may also associate with this like history of head injuries, depression, or hypertension. Like all types of dementia, Alzheimer's is also caused by brain cell death. Although AD is classified as a neurodegenerative dementia, considerable evidence links vascular dysfunction and vascular risk factors as pathogenesis of AD. However, it is a progressive brain cell death that happens over a course of time and treatments can't stop Alzheimer's from progressing, they can temporarily slow the worsening of dementia symptoms and improve quality of life for those with Alzheimer's and their caregivers (www.alz.org; www.who.int).

Sovateltide is an endothelin B (ETB) receptor agonist (previously used names IRL-1620, SPI-1620 and PMZ-1620; International Non-proprietary Name (INN) approved by WHO is sovateltide). Activation of ETB receptors with PMZ-1620 produces neurovascular repair and remodeling or neuroregeneration. There are hidden stem cells in the brain, which becomes active following injury to the brain. Intravenous administration of PMZ-1620 (sovateltide) augments the activity of neuronal progenitor cells in the brain to repair the damage by formation of new mature neurons and blood vessels. In addition, PMZ-1620 has anti-apoptotic activity and also increases cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females Aged 45 years through 85 years (have not had their 86th birthday)
2. Men and women with a diagnosis of Alzheimer's disease according to the clinical criteria
3. Women must be of non-childbearing potential, surgically sterile, or willing to use adequate birth control; men who are sexually active will also be required to use adequate birth control
4. Able to give consent for participation on their own or through their Legally Acceptable Representative
5. MRI/CT scan assessment within six months before baseline, corroborating the clinical diagnosis of AD and excluding other potential causes of dementia, especially cerebrovascular lesions
6. MMSE score in between 11 to 26 in case of mild to moderate stage of Alzheimer's disease

6. Absence of major depressive disease according to Geriatric Depression Scale (GDS) of < 5 7. Previous decline in cognition for more than six months as documented in subject's medical records 8. Subject, who are on stable treatment with any of AD drugs are also eligible to participate in this study 9. Formal education for eight or more years 10. Subjects living at home or nursing home setting, without continuous nursing care 11. General health status acceptable for participation in a 6-months clinical trial 12. A caregiver available and living in the same household or interacting with the subject a sufficient time each week and available if necessary to assure administration of drug 13. Subjects with any other chronic conditions are stable and undergoing appropriate treatment

Exclusion Criteria:

1. Subjects who have a Mini Mental State Examination (MMSE) score of < 10
2. Subjects who have serious or unstable medical conditions that would exclude completion of all procedures and data collection for the study, or would be likely to preclude participation in a drug development trial
3. A current Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnosis of active major depression, schizophrenia or bipolar disorder
4. Other infectious, metabolic or systemic diseases affecting the central nervous system
5. Subjects who have participated in a clinical trial investigating an anti-amyloid agent
6. Subjects who are currently participating in a clinical trial with an investigational drug
7. Subjects who, in the opinion of the physician, are otherwise unsuitable for this study
8. Clinically significant, advanced or unstable disease that may interfere with outcome measures, and which may bias the assessment of the clinical or mental status of the subject or put the subject at special risk
9. History of or screening brain MRI scan indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma)
10. Subject has had a myocardial infarction, unstable angina, stroke, transient ischemic attack or required intervention for any of these conditions within 6 months of Screening
11. Clinical or laboratory findings consistent with:

    1. Other primary degenerative dementia,
    2. Other neurodegenerative condition
    3. Seizure disorder
12. Subjects, who are already taking sedatives, antidepressants, antipsychotics and antihistaminic medications

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Incidence of PMZ-1620 related adverse events | 160 days
  The primary objective of the study is to determine incidence of drug (PMZ-1620) related adverse events.
Number of patients not receiving full treatment due to intolerance to PMZ-1620 | 160 days
  Tolerability will be determined by the number of patients that do not receive all the 18 doses of PMZ-1620.

SECONDARY OUTCOMES:
Changes in clinical progression of AD as measured by Mini-Mental State Examination (MMSE) | 160 days
  Statistically relevant changes in clinical progression of AD as measured by MMSE after 3 and 6 months of treatment. Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
Changes in neuropsychiatric inventory (NPI) Score | 160 days
  Statistically relevant changes in NPI Score after 3 and 6 months of treatment. The Neuropsychiatric Inventory (NPI) is designed to detect, quantify and track changes of psychiatric symptoms in a demented population. The NPI examines 12 sub-domains of behavioral functioning: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances, and appetite and eating abnormalities. Maximum is 144 points, where less number of points is mild behavioral disturbance and more number of points is severe behavioral disturbance.
Changes in Alzheimer's disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | 160 days
  Statistically relevant changes in ADAS-Cog after 3 and 6 months of treatment. Alzheimer's disease Assessment Scale-Cognitive Subscale is a commonly used objective measure of cognitive change. It is designed to measure cognitive areas commonly seen to decline in AD patients.Total scores range from 0-70, with higher scores indicating greater cognitive impairment. Many regulatory authorities recognize a four-point change on the ADAS-Cog at 6 months as indicating a clinically important difference.
Changes in hippocampal atrophy using MRI/CT | 160 days
  Changes in hippocampal atrophy using MRI/CT before and at the end of study
Changes in electroencephalograms (EEGs) | 160 days
  Changes in electroencephalograms (EEGs) suggestive progression in AD symptom after 3 and 6 months of treatment. A decline of posterior slow-frequency alpha power which is peculiar feature of Alzheimer's disease and an amplitude increase of widespread delta and theta and an amplitude decrease of posterior alpha and/or beta sources that are reflective of Alzheimer's disease will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, Study Chair — Pharmazz, Inc.
Locations (5):
- India (5):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - King George's Medical University, Lucknow
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Seth GSMC & KEM Hospital, Mumbai
  - All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: No
Results will be communicated and published as manuscript

REFERENCES:
- [Background] Gulati A, Hornick MG, Briyal S, Lavhale MS. A novel neuroregenerative approach using ET(B) receptor agonist, IRL-1620, to treat CNS disorders. Physiol Res. 2018 Jun 27;67(Suppl 1):S95-S113. doi: 10.33549/physiolres.933859. PMID 29947531
- [Background] Briyal S, Nguyen C, Leonard M, Gulati A. Stimulation of endothelin B receptors by IRL-1620 decreases the progression of Alzheimer's disease. Neuroscience. 2015 Aug 20;301:1-11. doi: 10.1016/j.neuroscience.2015.05.044. Epub 2015 May 27. PMID 26022359
- [Background] Briyal S, Shepard C, Gulati A. Endothelin receptor type B agonist, IRL-1620, prevents beta amyloid (Abeta) induced oxidative stress and cognitive impairment in normal and diabetic rats. Pharmacol Biochem Behav. 2014 May;120:65-72. doi: 10.1016/j.pbb.2014.02.008. Epub 2014 Feb 20. PMID 24561065